CLINICAL TRIAL: NCT06516679
Title: Efficacy of Risk-Stratified Treatment in Newly Diagnosed Infant Leukemia: A Multicenter, Prospective Study
Brief Title: Efficacy of Risk-Stratified Treatment in Newly Diagnosed Infant Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2023-1263
Record Dates: First submitted 2024-06-27; First posted 2024-07-24 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Leukemia, Lymphoid
MeSH Terms: conditions — Leukemia, Lymphoid

STUDY DESIGN:
Intervention Model Description: * Low risk group : KMT2A wild type & minimal residual disease(MRD) (-) after consolidation 1
  * Intermediate risk group : Intermediate risk (If one of the two cases below applies)
    * KMT2A: MLL mutation (+) & minimal residual disease (MRD) (-) after consolidation 1
      * KMT2A: wild type & minimal residual disease (MRD) (+) after consolidation 1
  * High risk group : Somatic KMT2A mutation (+) & minimal residual disease (MRD) (+) after consolidation 1
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low risk group (Experimental): KMT2A wild type & minimal residual disease(MRD) (-) after consolidation 1
  Interventions: Drug: Consolidation #4(without daunorubicin)
- Intermediate risk group (Experimental): ntermediate risk (If one of the two cases below applies)
  * KMT2A: MLL mutation (+) & minimal residual disease (MRD) (-) after consolidation 1
    * KMT2A: wild type & minimal residual disease (MRD) (+) after consolidation 1
  Interventions: Drug: Consolidation #4(with daunorubicin)
- High risk group (Experimental): Somatic KMT2A mutation (+) & minimal residual disease (MRD) (+) after consolidation 1
  Interventions: Drug: Allogeneic hematopoietic stem cell transplantation after Consolidation #4(with daunorubicin)

INTERVENTIONS:
Drug: Consolidation #4(without daunorubicin) — 1. Induction chemotherapy(5wks) : Prednisolone, Dexamethasone, Vincristine, Daunorubicin, L-asparaginase, Cytarabine, intrathecal cytarabine, intrathecal methotrexate
  2. Low Risk Cosolidation 1 chemotherapy(3wks) : Cytarabine, Etoposide, Cyclophosphamide, intrathecal methotrexate
  3. Low Risk Cosolidation 2 chemotherapy(3wks) : Methotrexate, 6-mercaptopurine, intrathecal methotrexate
  4. Low Risk Cosolidation 3 chemotherapy(3wks) : Cytarabine, L-asparaginase, intrathecal methotrexate
  5. Low Risk Cosolidation 3 chemotherapy(8wks) : Dexamethasone, Vincristine, Daunorubicin, Cytarabine, Cyclophosphamide, 6-mercaptopurine, intrathecal methotrexate
  6. Maintenance chemotherapy(about 2yrs) : Vincristine, Dexamethasone, 6-mercaptopurine, intrathecal methotrexate
  Arms: Low risk group
Drug: Consolidation #4(with daunorubicin) — 1. Induction chemotherapy(5wks) : Prednisolone, Dexamethasone, Vincristine, Daunorubicin, L-asparaginase, Cytarabine, intrathecal cytarabine, intrathecal methotrexate
  2. High Risk Cosolidation 1 chemotherapy(3wks) : Cytarabine, Etoposide, Cyclophosphamide, Daunorubicin intrathecal methotrexate
  3. High Risk Cosolidation 2 chemotherapy(3wks) : Methotrexate, 6-mercaptopurine, intrathecal methotrexate
  4. High Risk Cosolidation 3 chemotherapy(3wks) : Cytarabine, L-asparaginase, intrathecal methotrexate
  5. High Risk Cosolidation 3 chemotherapy(8wks) : Dexamethasone, Vincristine, Daunorubicin, Cytarabine, Cyclophosphamide, 6-mercaptopurine, intrathecal methotrexate
  6. Maintenance chemotherapy(about 2yrs) : Vincristine, Dexamethasone, 6-mercaptopurine, intrathecal methotrexate
  Arms: Intermediate risk group
Drug: Allogeneic hematopoietic stem cell transplantation after Consolidation #4(with daunorubicin) — 1. Induction chemotherapy(5wks) : Prednisolone, Dexamethasone, Vincristine, Daunorubicin, L-asparaginase, Cytarabine, intrathecal cytarabine, intrathecal methotrexate
  2. High Risk Cosolidation 1 chemotherapy(3wks) : Cytarabine, Etoposide, Cyclophosphamide, Daunorubicin intrathecal methotrexate
  3. High Risk Cosolidation 2 chemotherapy(3wks) : Methotrexate, 6-mercaptopurine, intrathecal methotrexate
  4. High Risk Cosolidation 3 chemotherapy(3wks) : Cytarabine, L-asparaginase, intrathecal methotrexate
  5. High Risk Cosolidation 3 chemotherapy(8wks) : Dexamethasone, Vincristine, Daunorubicin, Cytarabine, Cyclophosphamide, 6-mercaptopurine, intrathecal methotrexate
  6. Allogeneic hematopoietic stem cell transplantation
  Arms: High risk group

SUMMARY:
This clinical trial is an open-label, multicenter, prospective phase 2 clinical trial targeting pediatric leukemia patients of infant age. The goal is to improve survival rates by varying the presence or absence of chemotherapy and hematopoietic stem cell transplantation based on genetic characteristics at the time of diagnosis and minimal residual disease (MRD) values measured by various methods after treatment.

In addition, by clearly defining the patient group that requires hematopoietic stem cell transplantation, it is expected that the role of hematopoietic stem cell transplantation in infantile leukemia, for which there have been various guidelines for hematopoietic stem cell transplantation, can be confirmed. Additionally, due to the characteristics of infants, this study aim to identify long-term sequelae or prognosis related to treatment by prospectively collecting side effect data related to treatment during and after treatment.

DETAILED DESCRIPTION:
Infant leukemia patients are classified into low/intermediate/high risk groups and hematopoietic stem cell transplantation is performed after chemotherapy or chemotherapy as shown in the schema below.

* Low risk group : Induction chemotherapy-Low Risk Consolidation chemotherapy 1~4 - Maintenance chemotherapy
* Intermediate risk group : Induction chemotherapy-High Risk Consolidation chemotherapy 1~4 - Maintenance chemotherapy
* High risk group : Induction chemotherapy-High Risk Consolidation chemotherapy 1~4 - hematopoietic stem cell transplantation

ELIGIBILITY:
Inclusion Criteria:

* The age of diagnosis is less than 1 year old
* The disgnosisi of ALL or ALAL(lymphoid predominant)
* Informed consent of the parents(guardians) before participation in this study

Exclusion Criteria:

* Burkitt leukemia/lymphoma or mature B-cell leukemia
* Down syndrome, Bloom syndrome, ataxia-telangiectasia, Fanconi anemia, Kostmann syndrome, Shwachman syndrome or other bone marrow failure syndrome, hematopoietic stem cell transplantation
* Relapsed infant leukemia
* Participants with contraindication to medication
* Administered systemic steroid therapy within 4 weeks prior to this study
* Participants in other interventional studies other than this protocol

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2032-08-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
3-years Overall survival(OS) rate | 3-years
  The 3-years overall survival rate defined as the percentage of subject in a treatment group who are alive three years after the start of treatm

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 5years
  The overall survival rate defined as the percentage of subject in a treatment group who are alive five years after the start of treatment.
Event Free Survial(EFS) | 3-years and 5-years
  EFS is defined as the period from study enrollment until disease progression, including hematological recurrence of ALL, development of secondary malignancy, or death from any causes, whichever occurs earlier.
The rate of hematopoietic stem cell transplant patients by risk group | Up to 5years
  through study completion, an average of 1 year
recurred rate | Up to 5years
  As a the period from enrollment to disease progression/recurrence
Death rate related to infusion | Up to 5years
  The time until defined by date of drug-related mortality from the date of 1st infusion

CONTACTS AND LOCATIONS:
Locations (8):
- South Korea (8):
  - Chonnam National University Hwasun Hospital, Hwasun
  - Jeju National University Hospital, Jeju City
  - Pusan National University Yangsan Hospital, Pusan
  - Asan Medical Center, Seoul
  - Samsung Medical Cente, Seoul
  - Seoul National University Hospital, Seoul
  - Seoul saint Mary's Hospital, Seoul
  - Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No